CLINICAL TRIAL: NCT03048578
Title: Clinical Efficacy and Safety of Using 3.0mg Liraglutide to Treat Weight Regain After Roux-en-Y Gastric Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-01527
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Obesity
Keywords: Roux-en-Y gastric bypass (RYGB)
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Randomization will be 2:1 (drug:placebo) with stratification by gender and percent post-operative TBWL (25%, 25 - 49.9%).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saxenda (Experimental): Week 1: 0.6mg/day Week 2: 1.2mg/day Week 3: 1.8mg/day Week 4: 2.4mg/day Week 5 and Onward: 3.0mg/day
  Interventions: Drug: Saxenda
- Placebo (Placebo Comparator): Week 1: 0.6mg/day Week 2: 1.2mg/day Week 3: 1.8mg/day Week 4: 2.4mg/day Week 5 and Onward: 3.0mg/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxenda — Week 1: 0.6mg/day Week 2: 1.2mg/day Week 3: 1.8mg/day Week 4: 2.4mg/day Week 5 and Onward: 3.0mg/day
  Other Names: Victoza
  Arms: Saxenda
Drug: Placebo — Subcutaneous Saline Solution
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial of liraglutide versus placebo over a follow-up period of 12 months in patients at least 18 months following Roux-en-Y gastric bypass (RYGB) who are experiencing weight regain. This study will assess the efficacy of liraglutide in improving cardiometabolic risk profile (as indicated by serum lipids, HbA1c, and waist circumference) and quality of life (as assessed by PHQ-9 (Patient Health Questionnaire), versus placebo in patients at least 18 months following RYGB who are experiencing weight regain as well as the safety of liraglutide in this patient population.

DETAILED DESCRIPTION:
The specific aims of this study are to:

* To evaluate the effects of liraglutide on body weight loss in patients who are experiencing weight regain following RYGB.
* To evaluate the effects of liraglutide on cardiometabolic risk and quality of life in patients who are experiencing weight regain following RYGB.
* To evaluate the safety of liraglutide in post-RYGB subjects.
* To evaluate the changes in obesity-related comorbid conditions in patients who are experiencing weight regain following RYGB.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 months status-post RYGB
* BMI 27 kg/m2 or greater in the presence of at least one weight-related comorbid condition
* BMI 30 kg/m2 or greater
* Regain of ≥10% of maximum TBWL post-RYGB
* Ability to provide informed consent before any trial-related activities
* Express willingness to follow protocol requirements

Exclusion Criteria:

* Pregnancy at time of enrollment
* Intention of becoming pregnant or breast feeding in the next 12 months
* Females of childbearing potential who are not using adequate contraceptive methods
* Presence of acute psychiatric problems or immaturity which would compromise cooperation with the study protocol
* Presence of biliary disease
* Known or suspected allergy to liraglutide or any product components
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* History of pancreatitis
* History of alcoholism
* History of Type 1 DM (Diabetes Mellitus)
* History of previous bariatric surgery other than RYGB except h/o LAGB and band removal.
* >10 years status-post RYGB
* < 25% TBWL at post-RYGB weight nadir
* >50% post-operative TBWL at time of screening
* Simultaneous use of any weight loss medications
* Use of insulin at the time of enrollment
* Current use of any GLP-1 agonist medication
* History of taking any GLP-1 agonist medication
* Participation in another ongoing clinical study
* Conditions that, in the opinion of the principal investigator, may jeopardize the patient's well-being and/or the soundness of this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Lofton, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saxenda | Placebo
Started | 89 | 43
Completed | 58 | 23
Not Completed | 31 | 20
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 22 | 10
Not completed — Adverse Event | 1 | 2
Not completed — Terminated | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxenda | Placebo | Total
Number analyzed (Participants) | 58 | 23 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (8.9) | 50.4 (11.9) | 49.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 20 | 69
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 50 | 20 | 70
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 15 | 8 | 23
  White | 32 | 13 | 45
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 8 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 58 | 23 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Losing at Least 5% Enrollment Body Weight Measured Using Cochran-Mantel-Haenszel (CMH) Test
Description: CMH is a test used in the analysis of stratified or matched categorical data. It allows testing of the association between a binary predictor or treatment and a binary outcome such as case or control status while taking into account the stratification
Time Frame: 12 Months
Measure: Number; unit: percentage of participants
Arm/Group | Saxenda | Placebo
Number analyzed (Participants) | 58 | 23
percentage of participants | 76 | 17

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Saxenda | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/43
Serious Adverse Events (participants affected / at risk) | 4/89 | 6/43
Other Adverse Events (participants affected / at risk) | 40/89 | 26/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxenda (N=89) | Placebo (N=43)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
HEPATITIS A (Infections and infestations) | 1 | 0
INTERNAL HERNIA (Gastrointestinal disorders) | 1 | 0
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SURGERY (Surgical and medical procedures) | 1 | 1
SYNCOPE (General disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saxenda (N=89) | Placebo (N=43)
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 1
ABNORMAL KIDNEY FUNCTION (Renal and urinary disorders) | 1 | 0
ACID REFLUX (Gastrointestinal disorders) | 2 | 0
AGGRAVATED GERD (Gastrointestinal disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
BAD MOUTH TASTE (General disorders) | 1 | 0
BURNING SENSATION AT INJECTION S (Skin and subcutaneous tissue disorders) | 1 | 0
CHEST TIGHTNESS (General disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 14 | 4
DECREASED APPETITE (General disorders) | 4 | 0
DIARRHEA (Gastrointestinal disorders) | 4 | 3
DIZZINESS (General disorders) | 1 | 0
DRY MOUTH (General disorders) | 4 | 3
ED VISIT (Surgical and medical procedures) | 1 | 0
EXCESSIVE PERSPIRATION (General disorders) | 1 | 0
FATIGUE (General disorders) | 6 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 2
GASTRITIS (Gastrointestinal disorders) | 0 | 1
GOUT FLARE (Musculoskeletal and connective tissue disorders) | 1 | 0
HAIR LOSS (General disorders) | 0 | 1
HEADACHE (General disorders) | 7 | 1
HIGH BLOOD PRESSURE (Cardiac disorders) | 1 | 0
HIGH ENERGY (General disorders) | 1 | 2
INCREASED ALCOHOL CONSUMPTION (General disorders) | 0 | 1
INCREASED CREATININE (AGGRAVATED) (Renal and urinary disorders) | 1 | 0
INJECTION SITE SWELLING (Skin and subcutaneous tissue disorders) | 1 | 0
INSOMNIA (General disorders) | 3 | 2
LACK OF APPETITE (General disorders) | 2 | 0
MOOD CHANGES - INCREASED IRRITABI (Psychiatric disorders) | 0 | 1
MUSCLE SPASM (Musculoskeletal and connective tissue disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 21 | 3
NIGHTTIME BINGE EATING (Psychiatric disorders) | 0 | 1
PALPITATIONS (Cardiac disorders) | 1 | 0
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
REDNESS AT INJECTION SITE (Skin and subcutaneous tissue disorders) | 0 | 1
SENSITIVITY TO COLD (LIGHTHEADNES (General disorders) | 0 | 1
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STOMACH PAIN (Gastrointestinal disorders) | 1 | 0
SWOLLEN SALIVARY GLAND (Endocrine disorders) | 0 | 1
SWOLLEN THYROID GLAND (Endocrine disorders) | 0 | 1
TIGHT CHEST (General disorders) | 1 | 0
URGENCY TO URINATE (Renal and urinary disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03048578/Prot_SAP_000.pdf